CLINICAL TRIAL: NCT05681026
Title: Cultural Tailoring and Pilot Testing of an Inpatient Yoga Therapy Program for Cancer Patients Undergoing Hematopoietic Stem Cell Transplantation in India, Tanzania, and the United States
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0785; NCI-2022-10563 (Other: NCI-CTRP Clinical Trials Registry); 3P30CA016672-46S3 (NIH)
Record Dates: First submitted 2022-12-15; First posted 2023-01-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic Stem Cell Transplantation; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga Sessions (Experimental): Participants will take part in Yoga of gentle movements, breathing exercises, relaxation techniques, and meditation all tailored to the participant's needs.
  Interventions: Behavioral: Yoga Sessions; Behavioral: Questionnaries; Behavioral: Interviews

INTERVENTIONS:
Behavioral: Yoga Sessions — Participants will have up to 12 sessions, 3 sessions per week starting two weeks before the transplant and throughout the first 30 days of your hospitalization.
Behavioral: Questionnaries — Participants will complete 4 questionnaires about any symptoms you may be having, any anxiety and/or depression you may be having, your quality of life, and your expectations about your treatment.
Behavioral: Interviews — Participants will have an exit interview last about 30-45 minutes. The interview will be conducted over the phone or remotely over Zoom, FaceTime, or other approved video call methods.). The interview will be audio and video recorded and transcribed (typed).

SUMMARY:
To develop and measure the effects of a culturally sensitive yoga program for inpatients

DETAILED DESCRIPTION:
Primary Objective:

1. To develop a culturally tailored yoga therapy (YT) program for HSCT patients. We will conduct semi-structured interviews with patients from each center to examine cultural norms, culturally sensitive language, and specific factors relevant to yoga and psychosocial support.

Secondary Objectives:

1. To optimize the HSCT YT program using an iterative process. Fifteen patients from each center (or until thematic saturation based on exit interviews) will participate in the yoga program two weeks prior to the transplant and throughout the first 30 days of the HSCT. Sessions will be delivered in person, via telehealth (Zoom), or in combination.
2. To examine the feasibility of adherence and follow-up completion. We will declare the intervention feasible if: (a) at least 50% of patients complete a minimum of 50% of the 12 YT sessions, and (b) at least 60% of participants complete follow-up measures at 2 months after transplant (± 7 days).

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients scheduled to undergo an autologous or allogeneic HSCT at MD Anderson, HCG, or MNH;
2. Age 18 or older;
3. English, Hindi, or Swahili speaking;
4. Able to sign a written informed consent and be willing to follow protocol requirements.

Exclusion Criteria:

* Extreme mobility issues that preclude participating in the YT;
* Major thought disorders such as schizophrenia or uncontrolled bipolar disorder;
* HCT comorbidity score of 3 or higher, excluding cancer diagnoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-8 (PHQ-8) | through study completion; an average of 1 year
  The PHQ-8 is a 8-item self-report questionnaire used to assess bother of depressive symptoms over the past 2 weeks. The PHQ-8 is a 8-item questionnaire to screen for degree of depressive symptoms scored on a 0-24 scale with higher scores indicating greater distress and impairment

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- M D Anderson Cancer Center, Houston, Texas, United States
- Swami Vivekananda Yoga Anusandhana Samsthana, Giddenahalli, Karnataka, India
- Muhimbili National Hospital, Dar es Salaam, Tanzania

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org